CLINICAL TRIAL: NCT00333671
Title: Diabetic Macular Oedema: the Retinal Thickness as a Function of Changes in Plasma Osmolality Evaluated by OCT.
Brief Title: Quantification of Rising the Osmotic Pressure in Diabetic Intraretinal Fluid Accumulation (Diabetic Macular Oedema)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Birgit Sander, Principal Investigator, Glostrup University Hospital, Copenhagen
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Dorte Nellemann, glycerol
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Macular Oedema
Keywords: Macular oedema; Diabetes; Pathogenesis; Osmolality; Retinal thickness
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus | interventions — Glycerol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Glycerol

SUMMARY:
Diabetic macular oedema is characterized by fluid accumulation in the retinal tissue from leaking retinal vessels, the capillaries. This state can lead to severe visual loss and blindness. According to basic physiologic rules several factors influence the fluid transport between the capillaries and the surrounding tissue. One of these factors is the balance between the large molecules within the vessel lumen and the retinal tissue. Some drugs change this balance, the osmotic balance, by moving the fluid from the tissue to the vessel lumen. In relation to diabetic macular oedema, treatment with such a drug potentially would reduce the retinal thickness because it extracts fluid from the retinal tissue. Glycerol has this potential. If reduction of the thickness with glycerol is confirmed, then it proves the significance of the osmotic balance in the basic nature of diabetic macular oedema.

In this study we therefore examine the time dependent change in retinal thickness after glycerol intake by an instrument called optical coherence tomography (OCT). The participants drink glycerol and the thickness of the retina is then monitored closely by OCT during the following three hours. Since diabetic changes in the retina are focal pr. definition, the secondary purpose of the study is to find any regional differences in the response. The examinations are repeated at a second visit where the patient drink another dose of glycerol, because we also want to analyse for a dose dependent response. Which dose is given at each visit is randomised on beforehand. In addition to measuring the retinal thickness a variety of examinations are performed both before and during the study, e.g. blood samples and systemic blood pressure measurements.

DETAILED DESCRIPTION:
In general, when oedema is present, increasing the osmotic pressure in the retinal capillaries by an osmotic drug induces transcapillary fluid transport from the retinal tissue to the vascular lumen, according to the Starling equation. Theoretically, in diabetic macular oedema the event would lead to reduction of the retinal thickness, which could then be visualised by Optical Coherence Tomography. The main purpose of this trial is therefore to evaluate and quantify the changes in retinal thickness of the oedema after increasing the intracapillary osmotic pressure with glycerol ingestion. A reduction of the retinal thickness will confirm the application of the Starling osmotic forces on diabetic macular oedema. Secondly, we want to describe any regional differences in the retinal response and analyse for dose dependent variations.

Principles of material and methods: A prospective, randomized, clinical trial on 15 patients with diabetic significant macular oedema. At baseline the patients undergo a thorough ophthalmologic examination including ETDRS visual acuity, slit lamp biomicroscopy, Optical Coherence Tomography (Stratus-OCT), 7-field fundus photography followed by fluorescein angiography. In addition the systemic blood pressure is measured and blood samples are taken to rule out severe renal insufficiency and to estimate glycosylated haemoglobin.

The patients are all randomised to drink either 1.5 or 3 mL glycerol/kg body weight (max. 250 mL pr day) on the first of two visit dates. The last dose is given at the second visit. In the following three hours the retinal thickness is then monitored closely by Stratus-OCT after the glycerol ingestion.

The plasma osmolality and plasma triglyceride (an indirect indicator of glycerol) are confirmed by venous blood samples, also at predetermined times after the last swallow of glycerol. In addition the systemic blood pressure and the capillary blood glucose are monitored closely during the visit.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic significant macular oedema (by biomicroscopy or OCT)
* Visual acuity of minimum 60 letters by the ETDRS chart (4 m distance)
* ETDRS grade between 35 and 53, both stages included
* baseline blood pressure of max. 160/90 mmHg
* informed consent

Exclusion Criteria:

* another macular disease than diabetic macular oedema to explain the symptoms, incl. prior laser photocoagulation
* pregnancy
* moderate to severe heart or lung disease (crural oedemas, dyspnoea during low activity, or basal crackles by lung stethoscopy
* renal insufficiency with albumin excretion larger than 300 g/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-12; Primary Completion 2006-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Retinal thickness by fast retinal thickness mapping by optical coherence tomography at times 0, 2, 4, 8, 10, 15, 20, 30, 60, 90, 120 and 180 minutes after the last swallow of glycerol.

SECONDARY OUTCOMES:
Regional differences in response by fast retinal thickness mapping by optical coherence tomography at times 0, 2, 4, 8, 10, 15, 20, 30, 60, 90, 120 and 180 minutes after the last swallow of glycerol
dose dependent differences in the same time spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Nellemann Thornit, MD, Principal Investigator — Department of Ophthalmology, Glostrup Hospital, University of Copenhagen, Nordre Ringvej 57, DK-2600 Glostrup, Denmark
Locations (1):
- Department of Ophthalmology, Herlev Hospital, University of Copenhagen, Herlev Ringvej 75, Herlev, Denmark

REFERENCES:
- [Derived] Thornit DN, Vinten CM, Sander B, Lund-Andersen H, la Cour M. Blood-retinal barrier glycerol permeability in diabetic macular edema and healthy eyes: estimations from macular volume changes after peroral glycerol. Invest Ophthalmol Vis Sci. 2010 Jun;51(6):2827-34. doi: 10.1167/iovs.09-4172. Epub 2009 Dec 30. PMID 20042642